CLINICAL TRIAL: NCT06648772
Title: A Multicenter, Randomized, Double-blind, Vehicle-controlled Phase 3 Clinical Study To Evaluate The Efficacy and Safety Of Roflumilast Cream 0.3% (Zoryve®) in the Treatment of Plaque Psoriasis In China
Brief Title: Efficacy and Safety of Roflumilast Cream 0.3% in Subjects With Plaque Psoriasis: a Phase 3 Study
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HDM3014-301
Record Dates: First submitted 2024-10-09; First posted 2024-10-18 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-10

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Roflumilast Cream 0.3% (Experimental): For topical use, Q.D.
  Interventions: Drug: Roflumilast Cream 0.3%
- Vehicle cream (Placebo Comparator): For topical use, Q.D.
  Interventions: Drug: Vehicle cream

INTERVENTIONS:
Drug: Roflumilast Cream 0.3% — Roflumilast Cream 0.3%
  Other Names: Zoryve
  Arms: Roflumilast Cream 0.3%
Drug: Vehicle cream — Vehicle cream
  Arms: Vehicle cream

SUMMARY:
This study is a multi-center, randomized, double-blind, vehicle-controlled phase III study to evaluate the efficacy, safety, and PK profile of roflumilast cream 0.3% in Chinese subjects ≥6 years of age with plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the objectives and requirements of this study, voluntarily participate in the clinical trial and sign the informed consent form (ICF), and be able to complete all visits as required by the protocol.
2. Aged ≥ 6 years at the time of signing the ICF, male or female.
3. Clinical diagnosis of plaque psoriasis before the first dose in this study, with a disease duration of ≥ 6 months (for those aged ≥ 12 years) or ≥ 3 months (for those aged 6-11 years) and stable for the last 4 weeks.
4. Patients are required to meet the following requirements at screening and baseline:

   * Psoriasis involving 2%-20% BSA (excluding the scalp, palms, and soles);
   * IGA score of ≥ 2 points;
   * PASI score of ≥ 2 points (excluding the scalp, palms, and soles).
5. Females of childbearing potential (FOCBP) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test at Baseline. FOCBP must agree to take at least one reliable form of birth control, including oral/implantable/injectable/transdermal contraceptive, intrauterine device, bilateral tubal ligation/occlusion, partner's vasectomy, and barrier contraception (used correctly throughout sexual intercourse), from 4 weeks before the first dose of the IMP until 2 months after the last dose. If the subject is routinely abstinent, the subject may use this form of contraception, but should choose a reliable form of contraception as mentioned above if the subject is no longer abstinent. Male subjects will be required to have no plans to have children, no plans to donate sperm, and agree to use highly effective contraception. from the first dose of the investigational medicinal product until 4 months after the last dose.

   Note: FOCBP are defined as female subjects who have experienced menarche, have not reached a postmenopausal state (amenorrhea for at least 12 consecutive months, with no clear cause other than menopause and confirmd by FSH), and have no surgical (i.e., bilateral oophorectomy and/or bilateral salpingectomy and/or hysterectomy) or investigator-determined causes of permanent infertility (e.g., mullerian agenesis, etc.).
6. Subjects were assessed by the investigator to be free of other medical conditions that would interfere with the assessment of safety and efficacy based on medical history, physical examination, routine blood, blood biochemistry, urine, and other laboratory tests.

Exclusion Criteria:

1. Non-plaque psoriasis (e.g., guttate psoriasis, pustular psoriasis, erythrodermic psoriasis, and arthropathic psoriasis) or drug-induced psoriasis.
2. Skin disorders or other conditions that, in the judgment of the investigator, may interfere with the assessment of endpoints relevant to this study, including but not limited to: viral lesions, fungal and bacterial skin infections, parasitic infections, syphilis or tuberculosis-related skin manifestations, etc.
3. Prior use of etanercept within 4 weeks before the first dose of this study, or use of adalimumab and/or infliximab within 8 weeks before the first dose of this study, or prior use of another biologic within 12 weeks before the first dose of this study (or within 5 half-lives of the biologic at the time of the first dose of this study, whichever is longer).
4. Prior use of systemic drugs for psoriasis treatment or any other agents which may impact efficacy assessment of psoriasis, including but not limited to oral or intravenous glucocorticoids, retinoic acids, methotrexate, cyclosporine, and other systemic immunosuppressive agents or a class of drugs (including Chinese herbal formulas, herbs, proprietary Chinese medicines, etc.) containing Chinese medicinal ingredients within 4 weeks of the first dose of this study.
5. Prior use of topical agents for psoriasis treatment or any other agents which may impact efficacy assessment of psoriasis, including but not limited to topical glucocorticoids, vitamin D analogues, benvitimod and prescription emollients or emollients containing additives (e.g., ceramides, hyaluronic acid, urea, or filamentous proteolytic products) or antipruritic ingredients (e.g., menthol, polyhydroxyethanol, pramoxine, lidocaine, prilocaine, capsaicin, naltrexone, N-palmitoylethanolamine, etc.) or a class of drugs (including Chinese herbal formulas, herbs, proprietary Chinese medicines, etc.) containing Chinese medicinal ingredients for topical use (Note: for the treatment of diseases other than psoriasis, except in cases where the use of such medicines is deemed necessary in the medical judgment of the investigator and/or the specialist and would not interfere with the assessment of the study), etc. within 2 weeks.
6. Prior use of psoralen plus ultraviolet A (PUVA) or ultraviolet B (UVB) phototherapy within 4 weeks before the first dose of this study.
7. Prior use of ZORYVE® cream or foam; prior use of oral roflumilast or other phosphodiesterase-4 (PDE4) inhibitors (apremilast, etc.) within 4 weeks prior to the first dose of this study.
8. Prior use of antihistamines, potent cytochrome P (CYP) 450 enzyme inhibitors (such as indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone, saquinavir and telithromycin) or inducers (such as efavirenz, barbiturates, phenytoin sodium, and rifampicin) within 2 weeks before the first dose of this study or these drugs cannot be discontinued during the study.
9. Prior use of lithium-containing agents or antimalarials within 4 weeks (or 5 half-lives, whichever is longer) prior to the first dose of this study..
10. Subjects who are expected to have excessive exposure to natural/artificial light, sunbeds, or other light-emitting diode (LED) irradiation at the treatment area during the treatment period of this study.
11. Planned initiation or change in the use of an existing medication (e.g., beta-blockers or angiotensin-converting enzyme inhibitors) that, in the opinion of the investigator, can affect the efficacy evaluation for psoriasis.
12. Known hypersensitivity to roflumilast or any of the excipients of the product (white vaseline, isopropyl palmitate, hydroxybenzyl ester, propyl hydroxybenzoate, diethyleneglycol monoethyl ether, hexanediol, hydrochloric acid dilute, sodium hydroxide, Crodafos CES [including cetearyl alcohol, cetyl phosphate, and ceteareth-10 phosphate]).
13. Previous or suspected human immunodeficiency virus (HIV) infection, or HIV antibody-positive at screening; or hepatitis B (hepatitis B virus surface antigen [HBsAg])-positive or HBsAg-negative but hepatitis B virus core antibody (HBcAb)-positive, in which case DNA quantitation should be detected and the result is higher than the upper limit of normal; or hepatitis C (hepatitis C virus [HCV]) antibody-positive with HCV-RNA quantification above the upper limit of normal value; or syphilis screening-positive (except for patients with a positive specific antibody test, a negative non-specific antibody test, and confirmed as inactive infection in combination with clinical judgment).
14. As judged by the investigator, with known or suspected:

    * Moderate to severe hepatic impairment (Child-Pugh B/C) at screening. See Appendix 16.7 for Child-Pugh grading criteria
    * Total bilirubin and or AST and or ALT > 1.5 x ULN at screening
    * SCr > 1.5 x ULN at screening
    * History of major depressive disorder, suicidality, or suicidal tendency suggested by the C-SSRS at baseline or screening.
15. PHQ-8 (adults) or modified PHQ-A (aged 12-17 years) ≥ 10 points, for children aged 6-11 years, investigators assessed the presence or risk of depression after communicating with their parents/guardians at baseline or screening.
16. Female subjects in the lactating period; or subjects who have a fertility plan during the study.
17. Alcohol (defined as >2 units of alcohol per day/>14 units of alcohol per week, with 1 unit of alcohol equivalent to 360 mL of beer or 45 mL of spirits with 40% alcohol content or 150 mL of wine) or drug abuse within 6 months before screening in this study.
18. Have undergone a major surgery within 4 weeks prior to the first dose of this study (for the definition of major surgery, refer to Level 3 and Level 4 surgeries specified in the "Measures for the Classification of Surgical Procedures in Medical Institutions" issued by the National Health Commission of the People's Republic of China on Dec. 6, 2022) or plan to undergo a major surgery during the study.
19. Cancer (except for non-melanoma skin cancer, localized prostate cancer, ductal carcinoma in situ, stage I uterine cancer, cervical carcinoma in situ, or breast carcinoma in situ that have been treated with curative therapy) within 5 years before the first dose of this study.
20. Prior active infection requiring the use of oral or intravenous antibiotics, antifungal or antiviral agents within 7 days before the first dose of this study.
21. Any serious disease or medical measure, physical or mental condition that, in the opinion of the investigator, will affect the subject's participation in the trial (including the use of IMP and participation in required study visits), or that, in the opinion of the investigator, will pose a significant risk or effect to the subject.
22. Family members involving staff from the clinical research organization, contract research organization (CRO, if applicable), or sponsor participated in the design or conduct of this study, or a family member has already been enrolled in this study.
23. Currently participating in any other interventional clinical trials; or participation in a pharmaceutical clinical trial within 3 months or 5 half-lives (whichever is longer) or any other interventional clinical trial within 3 months prior to the first dose of this study.
24. Other reasons judged by the investigator as inappropriate for enrollment in this study.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 189 (Estimated)
Dates: Start 2024-11-14 (Actual); Primary Completion 2025-06-28 (Estimated); Study Completion 2025-07-04 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects achieving IGA treatment success after 8 weeks of treatment | Baseline, week 8
  The IGA is a static evaluation of qualitative overall psoriasis severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4). Each grade is defined by a distinct and clinically relevant morphologic description that minimizes inter-observer variability. Treatment success is defined as an IGA score of 0 or 1 with an improvement of ≥ 2 points from baseline.

SECONDARY OUTCOMES:
Proportion of subjects achieving PASI-75 after 8 weeks of treatment. | Baseline, Week 8
  PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). Subjects achieving PASI-75 are those who achieve a 75% reduction in PASI from baseline.
Proportion of subjects achieving PASI-90 after 8 weeks of treatment. | Baseline, Week 8
  PASI combines the assessment of the severity of lesions and the area affected into a single score in the range 0 (no disease) to 72 (maximal disease). Subjects achieving PASI-90 are those who achieve a 90% reduction in PASI from baseline.
Time required to achieve PASI-50 from baseline. | Until week 8
  Time required to achieve PASI-50 (i.e., PASI reduction ≥ 50% from baseline) from baseline.
Proportion of subjects achieving IGA treatment success after 4 weeks of treatment. | Baseline, Week 4
  The IGA is a static evaluation of qualitative overall psoriasis severity. This global assessment scale is an ordinal scale with five severity grades (reported only in integers of 0 to 4). Each grade is defined by a distinct and clinically relevant morphologic description that minimizes inter-observer variability. Treatment success is defined as an IGA score of 0 or 1 with an improvement of ≥ 2 points from baseline.
Proportion of subjects with an I-IGA score ≥ 2 points at baseline achieving an I-IGA score of 0 or 1 and an improvement of ≥ 2 points from baseline after 8 weeks of treatment | Baseline, Week 8
  I-IGA means Intertriginous area IGA. For subjects with intertriginous area involvement of at least 'mild' severity by IGA (I-IGA≥2) at Baseline (using the IGA scale but evaluating intertriginous areas ONLY and NOT whole body involvement), an I-IGA will be recorded.
Proportion of subjects with an I-IGA score ≥ 2 points at baseline achieving an I-IGA score of "0" after 8 weeks of treatment | Baseline, Week 8
  I-IGA means Intertriginous area IGA. For subjects with intertriginous area involvement of at least 'mild' severity by IGA (I-IGA≥2) at Baseline (using the IGA scale but evaluating intertriginous areas ONLY and NOT whole body involvement), an I-IGA will be recorded.
Proportion of subjects with WI-NRS of ≥ 4 at baseline and a decrease in WI-NRS of ≥ 4 from baseline after 2, 4, and 8 weeks of treatment | Week 2, 4, 8
  WI-NRS (Worst Itch Numerical Rating Scale) assessments will be performed for subjects 12 years and older. The WI-NRS will be determined by asking the subject's assessment of worst itch over the past 24 hours. The scale is from '0 to 10' ("no itch" to "worst imaginable itch").
Changes from baseline in the score of DLQI (aged ≥ 17 years)/CDLQI (aged 6-16 years) after 4 and 8 weeks of treatment | Week 4, 8
  Dermatology Life Quality Index (DLQI) and Children's Dermatology Life Quality Index (CDLQI) will be performed to measure how much skin problem has affected subjects' life over the last week.
Changes from baseline in the total score of PSD (for adult subjects only) after 4 and 8 weeks of treatment | From baseline to Week 4 and 8
  Psoriasis Symptom Diary (PSD) will be used to assess the improvement in psoriasis symptom.
treatment emergence adverse events | Throughout the study
  Incidence, severity, and causal relationship of treatment emergence adverse events (TEAE), TEAEs leading to withdrawal and death.
Trough concentration (Ctrough) | week 2, 4, 6, 8
  Trough concentration of plasma roflumilast and its N-oxide

CONTACTS AND LOCATIONS:
Locations (31):
- China (31):
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - People's Hospital of Peking University, Beijing
  - Beijing Children's Hospital, Capital Medical University, Beijing
  - Beijing Tongren Hospital, Capital Medical University, Beijing
  - Children's Hospital of Hunan Province, Changsha
  - The Second Xiangya Hospital of Central South University, Changsha
  - Affiliated Hospital of Chengde Medical College, Chengde
  - Sichuan Provincial People's Hospital, Chengdu
  - The Second People's Hospital of Chengdu, Chengdu
  - Affiliated Hospital of Chongqing Three Gorges Medical College, Chongqing
  - The Second Affiliated Hospital of Chongqing Medical University, Chongqing
  - The Sixth People's Hospital of Dongguan, Dongguan
  - Enshi Tujia and Miao Autonomous Prefecture Central Hospital, Enshi
  - Dermatology Hospital of Southern Medical University, Guangzhou
  - Hainan Fifth People's Hospital, Haikou
  - The First People's Hospital of Hangzhou, Hangzhou
  - Zhejiang Provincial People's Hospital, Hangzhou
  - The Second Affiliated Hospital of Harbin Medical University, Harbin
  - Ji'nan Central Hospital, Ji'nan
  - The First Hospital of Jilin University, Jilin
  - The Fourth Affiliated Hospital of Zhejiang University School of Medicine, Jinhua
  - The Second Affiliated Hospital of Henan University of Science and Technology, Luoyang
  - Affiliated Hospital of Nantong University, Nantong
  - Sanmenxia Central Hospital, Sanmenxia
  - Shanghai Skin Disease Hospital, Shanghai
  - The Second Affiliated Hospital of South Anhui Medical College, Wuhu
  - The First Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - The First People's Hospital of Yancheng, Yancheng
  - Zhengzhou Central Hospital, Zhengzhou
  - Affiliated Hospital of Jiangsu University, Zhenjiang